CLINICAL TRIAL: NCT05021120
Title: A Phase 1a/1b, Multicenter, Open-Label, Dose-Escalation and Dose-Expansion Study to Evaluate the Safety, Pharmacokinetics, and Anti-tumour Activity of AK127 in Combination With AK104 in Subjects With Advanced or Metastatic Solid Tumours
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Antitumor Activity of AK127 in Combination With AK104 in Advanced and Metastatic Solid Tumours
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Akesobio Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Akeso (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK127-101
Record Dates: First submitted 2021-08-12; First posted 2021-08-25 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Advanced or Metastatic Solid Tumours

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Masking Description: None (open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/treatment (Experimental): Experimental
  Interventions: Drug: AK127; Drug: AK104

INTERVENTIONS:
Drug: AK127 — Subjects will receive AK127 by intravenous administration
Drug: AK104 — After AK127 infusion, on the same day subjects will receive AK104 by intravenous administration

SUMMARY:
A Phase 1 study to evaluate the safety, tolerability, PK, immunogenicity, pharmacodynamics, and preliminary antitumor activity of AK127 in combination with AK104.

DETAILED DESCRIPTION:
This is a , Phase 1, first-in-human, multicenter, open label, dose escalation and dose expansion study designed to evaluate the safety, tolerability, PK, immunogenicity, pharmacodynamics, and preliminary antitumor activity of AK127 in combination with AK104 in subjects with advanced and metastatic solid tumours. The study comprises of 2 phases: a dose escalation phase and a dose expansion phase. Dose escalation for AK127 will occur using the 3+3+3 model given with a fixed regimen of AK104. Dose expansion will open at the discretion of the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent
2. In Phase 1a, patients with relapsed or refractory advanced solid malignancies
3. In Phase 1b, patients must have received no more than three prior lines of systemic therapy
4. Subject must have at least one measurable lesion according to RECIST Version1.1.
5. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.
6. Available archived or fresh tumor tissue
7. Adequate organ function.
8. For dose-expansion cohorts (Phase 1b), subjects must be willing to provide two fresh biopsy samples (pre-treatment and on treatment), where clinically appropriate.
9. Females of childbearing potential and non-sterilized males who are sexually active must use an effective method of contraception from screening until 120 days after final dose of investigational product.

Exclusion Criteria:

1. History of severe hypersensitivity reactions to other mAbs.
2. Subjects with a condition requiring systemic treatment with either corticosteroid (> 10 mg daily ) or other immunosuppressive medications within 2 weeks of study drug administration.
3. Prior use of approved or investigational anti-TIGIT, anti-PVRIG, or anti-CD96 therapy
4. Receiving any Other anticancer therapy (e.g., chemotherapy, radiotherapy, biologic or hormonal therapy for cancer treatment. etc.) within 4 weeks prior to the first dose of treatment
5. Any major surgery within 4 weeks prior to the first dose of treatment
6. Receiving agents with immunomodulatory effect within 2 weeks prior to the first dose of treatment.
7. Active or prior documented inflammatory bowel disease
8. History of organ transplant.
9. History of interstitial lung disease, noninfectious pneumonitis except for those induced by radiation therapies.
10. Known active hepatitis B or C infections or history of HIV.
11. Receipt of live attenuated vaccines within 4 weeks prior to the first dose of investigational product.
12. Patients with severe heart and lung dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence and Nature of Adverse Events (AEs) | From the time of informed consent signed through to 90 days after end of treatment
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Number of participants with a Dose Limiting Toxicity (DLT) | Within the first six weeks of treatment
  DLTs will be assessed during the first treatment cycle and assessed as having a suspected relationship to study drug according to pre-specific criteria in the protocol.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Disease control rate (DCR) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with AK127 + AK104 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment until death due to any cause.
Area under the curve (AUC) of AK127+AK104 for assessment of pharmacokinetics | From first dose of treatment through to 90 days after end of treatment
  The endpoints for assessment of PK including serum concentrations of AK127+AK104 at different timepoints after treatment administration.
Maximum observed concentration (Cmax) of AK127 + AK104 | From first dose of treatment through to 90 days after end of treatment.
  The endpoints for assessment of PK of AK127+AK104 include serum concentrations of AK127+AK104 at different timepoints after treatment administration.
Minimum observed concentration (Cmin) of AK127+AK104 | From first dose of treatment through to 90 days after end of treatment
  The endpoints for assessment of PK of AK127+AK104 include serum concentrations of AK127+AK104 at different timepoints after treatment administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of treatment through to 90 days after end of treatment
  The immunogenicity of AK127+AK104 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Ashford Cancer Centre Research, Adelaide
  - Austin Health, Melbourne
  - Monash Health, Melbourne
  - Southside Cancer Care Centre, Sydney
  - The Kinghorn Cancer Centre, St Vincents Hospital Sydney, Sydney

IPD SHARING:
Plan to Share IPD: No